CLINICAL TRIAL: NCT02432794
Title: Prospective Randomized Clinical Trial on Delay Phenomenon Utility in Preventing Oesophagogastric Anastomotic Dehiscence After Ivor-Lewis Esophagectomy. Pilot Study.
Brief Title: Trial on Delay Phenomenon Utility in Preventing Anastomotic Leakage After an Esophagectomy
Acronym: APIL_2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Leandre Farran Teixidor, Chief of oesophagogastric surgery department, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APIL_2013
Record Dates: First submitted 2015-04-21; First posted 2015-05-04 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- delay phenomenon by arteriography (Experimental): intervention: delay phenomenon by arteriography. Patients who will be subjected a delay phenomenon by arteriographic procedure before esophageal resection surgery minimum 14 days before surgery.
  An angiogram of the celiac trunk is performed through a femoral access before and after the embolization. A 4-5 Fr Simmons or Cobra catheter is used for the catheterization and embolization of the left gastric artery, and 0.035-inch platinum coils are proximally placed from the main trunk in the splenic artery. When accessory left gastric arteries are present, they are catheterized and embolized as well. The right gastric artery catheterization is realized by a 4-5 Fr catheter and coils or microcoils are proximally placed in the artery as well.
  Interventions: Procedure: delay phenomenon by arteriographic approach
- control group (No Intervention): Patients who will be operated directly without gastric ischemic conditioning. The investigators don't performed any arteriography before the esophageal surgical resection

INTERVENTIONS:
Procedure: delay phenomenon by arteriographic approach — we improve the microvascularization of the gastric fundus occluding the right and left gastric artery, and splenic artery two weeks before surgery by arteriography
  Arms: delay phenomenon by arteriography

SUMMARY:
This is a randomized clinical trial to clarify if the delay phenomenon could reduce the incidence of oesophagogastric dehiscence after an esophagectomy for esophageal cancer comparing an experimental group vs control group. The delay phenomenon will be performed by an arteriographic approach.

DETAILED DESCRIPTION:
Subtotal esophagectomy with tubular gastroplasty to upper mediastinum and esophagogastric anastomosis (Ivor-Lewis procedure) is a very complex surgical technique. It is performed in patients with infracarinal esophageal carcinoma and is associated with a high morbidity rate in specialized centers (up to 60% in some groups). One of the most important postoperative complications is the oesophagogastric anastomotic leakage which leads to high morbidity (mediastinitis, respiratory failure, pleural effusion) and mortality rate (up to 60% depending on the reports).

The most important cause of anastomotic leakage is the stomach's extreme sensitivity to ischemic injury. There are several experimental studies that have demonstrated that the delay phenomenon before the esophageal resection surgery aims to improve blood perfusion after a period of time. Few studies, only case-reports, describe a decrease in the incidence of intrathoracic and cervical anastomotic leakage. May the delay phenomenon reduce the incidence of anastomotic intrathoracic leakage?. There aren't any prospective randomized controlled trials to answer this question.

For this reason the investigators propose to perform a prospective randomized controlled trial in patients who underwent a subtotal esophagectomy (Ivor-Lewis procedure), comparing two groups: one of them will be submitted to a delay phenomenon by arteriographic procedure before esophageal resection surgery, and the other one will be operated on directly, to demonstrate if the delay phenomenon can reduce the incidence of anastomotic esophagogastric leakage.

We decided to conduct this trial as a pilot study due to the fact that the number of patients needed to achieve statistical significance was to high and would have taken almost 10 years. We established a recruitment period of 3 years, in wich we intend to include 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring a subtotal esophagectomy with en-bloc resection and an intrathoracic esophagogastrostomy for esophageal cancer
* 18 or above years old
* Acceptance and signing the full informed consent

Exclusion Criteria:

* Absence of pancreatitis
* Anatomic vascular alteration that contraindicate the embolization (congenital celiac trunk stenosis, presence of arcuate ligament,etc,..)
* refuse to collaborate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | 7 days
  investigators will consider anastomotic dehiscence the presence of one or more of the following conditions: radiologic confirmation by water-soluble contrast study (gastrografin administered orally) or thoracoabdominal Tc with oral contrast of dehiscence of oesophagogastric anastomosis or the stapler end of the gastroplasty.
  When the clinical conditions of patient don't allow a Rx control investigators will consider an anastomotic leakage in these conditions:
  Thoracic drain output of oesophagogastric content with amylase > 40 ukAT/L, confirmation of anastomotic dehiscence by the surgeon during a reintervention, endoscopic confirmation of anastomotic leakage of the stapled end of the plasty and methylene blue output after oral administration (100 ml of water with 10ml of methylene blue)

SECONDARY OUTCOMES:
plasty ischemia | 7 days
  investigators will consider plasty ischemia when one or more of the following criteria is present:
  * endoscopic evidence of gastric mucosa ischemia
  * evidence of low captation of the plasty in a thoracoabdominal CT with endovenous contrast that requires a reintervention.
  * intraoperative mortality (during hospitalization and/or 30 days after surgery).
hospital stay | 90 days
  investigators will consider since the day of the surgery until the day the patient will be discharged from the hospital
major and minor morbidity | 90 days
  investigators will evaluate morbidity according to Clavien-Dindo classification
postoperative mortality | during hospitalization and/or 30 days after surgery
post-embolization morbidity | 30 days
  investigators will consider post-embolization morbidity the following situations:
  * abdominal pain with EVA>3 (evaluated by EVA classification )
  * pancreatitis diagnosed by abdominal pain and amylase > 5 uKat/L or by CT.
  * abscess, pseudocyst diagnosed by CT or during oesophageal surgery
  * spleen ischemia diagnosed by CT or abdominal ultrasound and needs some treatment
  * liver ischemia diagnosed by Ct or abdominal ultrasound
  * bleeding or artery dissection diagnosed during the embolization and needs some treatment
  * arterial pseudoaneurism diagnosed during the embolization or by CT
anastomotic stricture | 6 months
  investigators will consider anastomotic stricture when they observe a reduction of anastomotic diameter by oral contrast Rx and needs some treatment (endoscopic dilation or reintervention)

CONTACTS AND LOCATIONS:
Overall Officials: Leandre F Teixidor, Ph D, MD, Principal Investigator — Bellvitge University Hospital
Locations (1):
- Leandre Farran Teixidor, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Result] Gonzalez-Gonzalez JJ, Sanz-Alvarez L, Marques-Alvarez L, Navarrete-Guijosa F, Martinez-Rodriguez E. [Complications of surgical resection of esophageal cancer]. Cir Esp. 2006 Dec;80(6):349-60. doi: 10.1016/s0009-739x(06)70987-3. Spanish. PMID 17192218
- [Result] Schroder W, Beckurts KT, Stahler D, Stutzer H, Fischer JH, Holscher AH. Microcirculatory changes associated with gastric tube formation in the pig. Eur Surg Res. 2002 Nov-Dec;34(6):411-7. doi: 10.1159/000065709. PMID 12403940
- [Result] Farran Teixidor L, Llop Talaveron J, Galan Guzman M, Aranda Danso H, Miro Martin M, Bettonica Larranaga C, Estremiana Garcia F, Biondo S. [Surgical outcomes of esophageal cancer resection since the development of an Oesophagogastric Tumour Board]. Cir Esp. 2013 Oct;91(8):517-23. doi: 10.1016/j.ciresp.2012.12.005. Epub 2013 Apr 11. Spanish. PMID 23583091
- [Result] Patil PK, Patel SG, Mistry RC, Deshpande RK, Desai PB. Cancer of the esophagus: esophagogastric anastomotic leak--a retrospective study of predisposing factors. J Surg Oncol. 1992 Mar;49(3):163-7. doi: 10.1002/jso.2930490307. PMID 1548890
- [Result] Griffin SM, Shaw IH, Dresner SM. Early complications after Ivor Lewis subtotal esophagectomy with two-field lymphadenectomy: risk factors and management. J Am Coll Surg. 2002 Mar;194(3):285-97. doi: 10.1016/s1072-7515(01)01177-2. PMID 11893132
- [Result] Schroder W, Holscher AH, Bludau M, Vallbohmer D, Bollschweiler E, Gutschow C. Ivor-Lewis esophagectomy with and without laparoscopic conditioning of the gastric conduit. World J Surg. 2010 Apr;34(4):738-43. doi: 10.1007/s00268-010-0403-x. PMID 20098986
- [Result] Metzger R, Bollschweiler E, Vallbohmer D, Maish M, DeMeester TR, Holscher AH. High volume centers for esophagectomy: what is the number needed to achieve low postoperative mortality? Dis Esophagus. 2004;17(4):310-4. doi: 10.1111/j.1442-2050.2004.00431.x. PMID 15569369
- [Result] Liebermann-Meffert DM, Meier R, Siewert JR. Vascular anatomy of the gastric tube used for esophageal reconstruction. Ann Thorac Surg. 1992 Dec;54(6):1110-5. doi: 10.1016/0003-4975(92)90077-h. PMID 1449294
- [Result] Boyle NH, Pearce A, Hunter D, Owen WJ, Mason RC. Scanning laser Doppler flowmetry and intraluminal recirculating gas tonometry in the assessment of gastric and jejunal perfusion during oesophageal resection. Br J Surg. 1998 Oct;85(10):1407-11. doi: 10.1046/j.1365-2168.1998.00943.x. PMID 9782026
- [Result] Urschel JD. Ischemic conditioning of the rat stomach: implications for esophageal replacement with stomach. J Cardiovasc Surg (Torino). 1995 Apr;36(2):191-3. PMID 7790342
- [Result] Yuan Y, Duranceau A, Ferraro P, Martin J, Liberman M. Vascular conditioning of the stomach before esophageal reconstruction by gastric interposition. Dis Esophagus. 2012 Nov-Dec;25(8):740-9. doi: 10.1111/j.1442-2050.2011.01311.x. Epub 2012 Jan 31. PMID 22292613
- [Result] Akiyama S, Kodera Y, Sekiguchi H, Kasai Y, Kondo K, Ito K, Takagi H. Preoperative embolization therapy for esophageal operation. J Surg Oncol. 1998 Dec;69(4):219-23. doi: 10.1002/(sici)1096-9098(199812)69:43.0.co;2-7. PMID 9881938
- [Result] Isomura T, Itoh S, Endo T, Akiyama S, Maruyama K, Ishiguchi T, Ishigaki T, Takagi H. Efficacy of gastric blood supply redistribution by transarterial embolization: preoperative procedure to prevent postoperative anastomotic leaks following esophagoplasty for esophageal carcinoma. Cardiovasc Intervent Radiol. 1999 Mar-Apr;22(2):119-23. doi: 10.1007/s002709900346. PMID 10094991
- [Result] Lamas S, Azuara D, de Oca J, Sans M, Farran L, Alba E, Escalante E, Rafecas A. Time course of necrosis/apoptosis and neovascularization during experimental gastric conditioning. Dis Esophagus. 2008;21(4):370-6. doi: 10.1111/j.1442-2050.2007.00772.x. PMID 18477261
- [Result] Farran L, Miro M, Alba E, Bettonica C, Aranda H, Galan M, Rafecas A. Preoperative gastric conditioning in cervical gastroplasty. Dis Esophagus. 2011 May;24(4):205-10. doi: 10.1111/j.1442-2050.2010.01115.x. Epub 2010 Oct 11. PMID 21040153